CLINICAL TRIAL: NCT02710396
Title: Identifying Genetic Predictors of Durable Clinical Benefit to Pembrolizumab in Advanced Non-small Cell Lung Cancer (NSCLC) Alone and in Combination With Chemotherapy.
Brief Title: Genetic Predictors of Benefit to Pembrolizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Frontline pembrolizumab approved in NSCLC as monotherapy and in combination with chemotherapy representing a new standard of care.
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ5450; 1U54CA209997 (NIH); R01CA205426 (NIH)
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects will receive single agent pembrolizumab 200 mg IV will be administered every 3 weeks for up to 2 years.
  Interventions: Drug: Pembrolizumab
- Cohort 2 (Experimental): Subjects will receive pembrolizumab 200 mg IV every 3 weeks for up to 2 years with 2 cycles of nab-paclitaxel and carboplatin administered with cycles 1 and 2.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Nab-paclitaxel
- Cohort 3 (Experimental): Subject will receive pembrolizumab 200 mg IV every 3 weeks for up to 2 years with 2 cycles of pemetrexed and carboplatin administered with cycles 1 and 2.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2 (programmed cell death (PD) proteins).
  Pembrolizumab 200 mg will be administered IV every 3 weeks.
  Other Names: Keytruda; MK-3475; Lambrolizumab
Drug: Carboplatin — Carboplatin AUC (area under curve (AUC)) = 5 IV on day 1 every 3 weeks administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
  Other Names: Paraplatin
  Arms: Cohort 2; Cohort 3
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m2 IV on days 1, 8 and 15 every 3 weeks administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
  Other Names: Abraxane
  Arms: Cohort 2
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
  Other Names: Alimta
  Arms: Cohort 3

SUMMARY:
The primary objective is to determine if mutation load underlies sensitivity to pembrolizumab alone and in combination with chemotherapy. This will be a 3-arm, multi-center, open-label, non-randomized biomarker trial in patients with advanced, treatment-naive NSCLC. Patients will receive 1 of 3 possible cohorts as per investigator's discretion. Patients with non-squamous histology may receive any of the 3 cohorts; patients with squamous histology may receive either cohorts 1 and 2.

DETAILED DESCRIPTION:
Somatic mutations leading to cancer are related to endogenous or exogenous DNA damaging processes. The resultant mutations can be separated into two categories - (i) mutations that provide selective advantage for clonal expansion and (ii) mutations that do not result in growth advantage. The latter have been termed passenger mutations, while the former are referred to as driver mutations. It is widely believed that the number of driver mutations in a cancer sample is limited to a handful, usually two or more but less than ten. In contrast, the genome of a cancer can harbor more than a million somatic mutations most of which are considered to be passengers.

Several studies have shown that the passenger mutations may not be oncogenic drivers but may be of importance in adaptive immune resistance of a tumor. In particular the relevant mutations are likely to be the nonsynonymous exonic mutations in tumors; these may give rise to novel proteins that differ from their wild type counterparts and are immunogenically more relevant. The study will explore if there is a relationship between the genetic mutations and the success of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients of all histologies may enroll to Cohorts 1 and 2. Only patients of non-squamous histologies may enroll to Cohort 3. If enrollment to a cohort is completed, enrollment may continue to other open cohorts.
* Be willing and able to provide written informed consent/assent for the trial.
* Chemotherapy naïve NSCLC patients.For NSCLC patients with lung adenocarcinoma, tumors must be Epidermal Growth Factor Receptor (EGFR) and Anaplastic Lymphoma Kinase (ALK) wild-type; if a Kirsten Ras (KRAS) mutation is detected, EGFR and ALK testing is not required.
* Diagnosis must be documented by histology or cytology from brushings, washings, or needle aspiration of a defined lesion but not from sputum cytology.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Sufficient archived tumor material available (equivalent to 2 core biopsies or greater); if insufficient archived tumor material available new tumor biopsy is mandatory.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of treatment initiation.

  -- Hematological
* Absolute neutrophil count (ANC): ≥1,500 /mcL
* Platelets: ≥100,000 / microliter (mcL)
* Hemoglobin: ≥9 g/dL or ≥5.6 mmol/L

  -- Renal
* Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

  -- Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases

  -- Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C (HCV) RNA [qualitative] is detected).
* Has a known history of active tuberculosis (TB)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* History of allergy or hypersensitivity to any component of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Brahmer, J.R., et al., Clinical activity and safety of anti-PD1 (BMS-936558, MDX-1106) in patients with advanced non-small-cell lung cancer (NSCLC). J Clin Oncol, 2012(30): p. suppl; abstr 7509
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer JR. Harnessing the immune system for the treatment of non-small-cell lung cancer. J Clin Oncol. 2013 Mar 10;31(8):1021-8. doi: 10.1200/JCO.2012.45.8703. Epub 2013 Feb 11. PMID 23401435
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Matsushita H, Vesely MD, Koboldt DC, Rickert CG, Uppaluri R, Magrini VJ, Arthur CD, White JM, Chen YS, Shea LK, Hundal J, Wendl MC, Demeter R, Wylie T, Allison JP, Smyth MJ, Old LJ, Mardis ER, Schreiber RD. Cancer exome analysis reveals a T-cell-dependent mechanism of cancer immunoediting. Nature. 2012 Feb 8;482(7385):400-4. doi: 10.1038/nature10755. PMID 22318521
- [Background] DuPage M, Cheung AF, Mazumdar C, Winslow MM, Bronson R, Schmidt LM, Crowley D, Chen J, Jacks T. Endogenous T cell responses to antigens expressed in lung adenocarcinomas delay malignant tumor progression. Cancer Cell. 2011 Jan 18;19(1):72-85. doi: 10.1016/j.ccr.2010.11.011. PMID 21251614
- [Background] DuPage M, Mazumdar C, Schmidt LM, Cheung AF, Jacks T. Expression of tumour-specific antigens underlies cancer immunoediting. Nature. 2012 Feb 8;482(7385):405-9. doi: 10.1038/nature10803. PMID 22318517
- [Background] Castle JC, Kreiter S, Diekmann J, Lower M, van de Roemer N, de Graaf J, Selmi A, Diken M, Boegel S, Paret C, Koslowski M, Kuhn AN, Britten CM, Huber C, Tureci O, Sahin U. Exploiting the mutanome for tumor vaccination. Cancer Res. 2012 Mar 1;72(5):1081-91. doi: 10.1158/0008-5472.CAN-11-3722. Epub 2012 Jan 11. PMID 22237626
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects will receive single agent pembrolizumab 200 mg IV will be administered every 3 weeks for up to 2 years.
  Pembrolizumab: Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2 (programmed cell death (PD) proteins).
  Pembrolizumab 200 mg will be administered IV every 3 weeks.
- Cohort 2: Subjects will receive pembrolizumab 200 mg IV every 3 weeks for up to 2 years with 2 cycles of nab-paclitaxel and carboplatin administered with cycles 1 and 2.
  Pembrolizumab: Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2 (programmed cell death (PD) proteins).
  Pembrolizumab 200 mg will be administered IV every 3 weeks.
  Carboplatin: Carboplatin AUC (area under curve (AUC)) = 5 IV on day 1 every 3 weeks administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
  Nab-paclitaxel: Nab-paclitaxel 100 mg/m2 IV on days 1, 8 and 15 every 3 weeks administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
- Cohort 3: Subject will receive pembrolizumab 200 mg IV every 3 weeks for up to 2 years with 2 cycles of pemetrexed and carboplatin administered with cycles 1 and 2.
  Pembrolizumab: Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2 (programmed cell death (PD) proteins).
  Pembrolizumab 200 mg will be administered IV every 3 weeks.
  Carboplatin: Carboplatin AUC (area under curve (AUC)) = 5 IV on day 1 every 3 weeks administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
  Pemetrexed: Pemetrexed 500 mg/m2 IV administered for 2 cycles concurrently with cycles 1 and 2 of pembrolizumab.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 14 | 5 | 0
Completed | 14 | 5 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects enrolled to cohort 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 14 | 5 | 0 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 0 | 4
  >=65 years | 13 | 2 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 0 | 8
  Male | 8 | 3 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 3 | 0 | 12
  More than one race | 4 | 2 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 5 |  | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With NSCLC Who Achieved DCB
Description: Objective response to study treatment will be assessed by RECIST 1.1 by a study radiologist. Partial and complete responses will be confirmed by a repeat imaging occurring at least 4 weeks after the initial identification of response; unconfirmed responses will be considered stable or progressive disease dependent on results of the second CT scan. Durable clinical benefit (DCB) will be defined as stable disease (Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study), OR complete response (disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.), OR partial response (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) lasting longer than 6 months.
Time Frame: Up to 2 years
Population: Zero analyzed in Cohort 3 as zero subjects participated in Cohort 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 14 | 5 | 0
Participants | 3 | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as participants with a partial (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) or complete response (Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) as assessed by RECIST 1.1 criteria.
Time Frame: Up to 2 years
Population: Zero analyzed in Cohort 3 as zero subjects participated in Cohort 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 14 | 5 | 0
Participants | 4 | 1 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The length of time from treatment initiation to progression of disease (at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression) as assessed by RECIST 1.1.
Time Frame: Up to 2 years
Population: Zero analyzed in Cohort 3 as zero subjects participated in Cohort 3.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 14 | 5 | 0
months | 4.80 [1.61 to 11.53] | 3.94 [1.38 to 23.49] |

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment to death.
Time Frame: Up to 28 months
Population: Zero analyzed in Cohort 3 as zero subjects participated in Cohort 3.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 14 | 5 | 0
Months | 14.06 [5.95 to 20.37] | 23.49 [1.38 to 27.63] |

ADVERSE EVENTS:
Time Frame: Up to 28 months
Description: Zero subjects participated in Cohort 3.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 12/14 | 4/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 10/14 | 5/5 | 0/0
Other Adverse Events (participants affected / at risk) | 13/14 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=5) | Cohort 3 (N=0)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=5) | Cohort 3 (N=0)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Creatine phosphokinase Increase (Investigations) | 1 | 1 | 0
Creatinine Increased (Investigations) | 2 | 3 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 0
Fever (General disorders) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
International normalized ratio (INR) Increase (Investigations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 0
Pain (General disorders) | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 0
Platelet count decreased (Investigations) | 3 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infections and infestations (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT02710396/Prot_SAP_000.pdf